CLINICAL TRIAL: NCT02301286
Title: A Phase III Double-blind Placebo-controlled Randomised Trial of Aspirin on Recurrence and Survival in Colon Cancer Patients
Brief Title: A Trial of Aspirin on Recurrence and Survival in Colon Cancer Patients
Acronym: ASPIRIN
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Leiden University (Other)
Collaborators: Stichting voor Patienten met Kanker aan het Spijsverteringskanaal (SPKS) (Unknown); Dutch Colorectal Cancer Group (Other); Stichting Geriatrische Oncologie Nederland (GeriOnNe) (Unknown); Fonds NutsOhra (Other); Innovatiefonds Zorgverzekeraars (Other)
Responsible Party: Principal Investigator, GJLiefers, Surgical Oncologist, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P14.152
Record Dates: First submitted 2014-11-07; First posted 2014-11-25 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Colon Cancer; Adjuvant Therapy
Keywords: Acetylsalicylic acid; Colon cancer; Survival
MeSH Terms: conditions — Colonic Neoplasms | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin (Experimental): Patients treated with acetylsalicylic acid 80 mg once daily for 5 years. Patients will be stratified according to the admission of adjuvant chemotherapy.
  Interventions: Drug: Acetylsalicylic acid
- Placebo (Placebo Comparator): Patients treated with placebo. Patients will be stratified according to the admission of adjuvant chemotherapy.
  Interventions: Drug: Placebo Acetylsalicylic acid

INTERVENTIONS:
Drug: Acetylsalicylic acid
  Other Names: Aspirin
  Arms: Aspirin
Drug: Placebo Acetylsalicylic acid
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether acetylsalicylic acidis effective on the recurrence and survival of colon cancer patients.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effect of 80mg acetylsalicylic acid (given orally once daily for 5 years) on 5 year overall survival (OS) for stage II and III colon cancer patients of 45 years of age and older. Preclinical, epidemiologic and clinical evidence suggest that acetylsalicylic acid use may reduce overall cancer risk and mortality in colon cancer patients. It is a phase III double blind placebo controlled, randomized trial of adjuvant low-dose acetylsalicylic acid in colon cancer patients. Patients will be stratified at randomization by centre, age (<70 and ≥70 years) chemotherapy use (any versus none) and disease stage.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥45 years
* Patients must have TNM stage that is one of the following: pT3-4; N0-2 and M0, or pT1-2 and N1-2 (UICC stage II and III) (in case of >1 tumour: largest tumour is stage II or III)
* Patients must have completed surgical resection (R0) (both laparoscopic and open surgery) within 12 weeks of randomisation

Exclusion Criteria:

* Patients with rectal cancer (defined as tumour within 15 cm from the anal verge)
* Patients currently taking oral anti-coagulants or use of LMWH
* Patients currently taking acetylsalicylic acid for any reason
* Patients with a history of bleeding disorders or active gastric or duodenal ulcers
* Patients currently taking high dose systemic glucocorticoids.(≥ 30 mg predniso(lo)n)
* Patients with (suspected) (non-) polyposis syndrome (FAP/AFAP, MAP, Lynch syndrome)
* Patients with >100 polyps of the colon or a known hereditary syndrome of the colon in a first degree family member
* Allergy or intolerance to salicylates.
* Patients with a history of other malignancies in the last 5 years, except for SCC or CIN.
* Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
5 year overall survival | 5 years
  The time to an event for OS is defined as the time interval between the date of randomisation and the date of death.

SECONDARY OUTCOMES:
Disease Free Survival | 5 years
  The time to an event for DFS is defined as the time interval between the date of randomisation and the date of disease recurrence or death, whichever comes first. Recurrence of a disease can be a loco-regional recurrence, a distant recurrence or a new primary colon cancer. The evidence for recurrence must be documented in the patients' file.
Time to Treatment Failure | 5 years
  The time elapsed between randomisation until treatment discontinuation due to disease progression, unacceptable toxicity, death or any other event of interest.

CONTACTS AND LOCATIONS:
Overall Officials: G.J. Liefers, MD PhD, Principal Investigator — Leiden University Medical Center; J.E.A. Portielje, Professor, Principal Investigator — Leiden University Medical Center; R. Fodde, Professor, Principal Investigator — Erasmus Medisch Centrum
Locations (32):
- Netherlands (32):
  - Ziekenhuisgroep Twente, Almelo
  - Meander MC, Amersfoort
  - Wilhelmina Ziekenhuis, Assen
  - Amphia Ziekenhuis, Breda
  - IJsselland Ziekenhuis, Capelle aan den IJssel
  - Reinier de Graaf Gasthuis, Delft
  - Deventer Ziekenhuis, Deventer
  - Slingeland Ziekenhuis, Doetinchem
  - NijSmellinghe, Drachten
  - Ziekenhuis Gelderse Vallei, Ede
  - Catharina Ziekenhuis, Eindhoven
  - Maxima MC, Eindhoven
  - MST, Enschede
  - Admiraal de Ruijter Ziekenhuis, Goes
  - Beatrix Ziekenhuis, Gorinchem
  - Groene Hart Ziekenhuis, Gouda
  - Ziekenhuis St. Jansdal, Harderwijk
  - Elkerliek Ziekenhuis, Helmond
  - Spaarne Gasthuis, Hoofddorp
  - Leiden University Medical Center, Leiden
  - Alrijne Ziekenhuis, Leiderdorp
  - HMC, Leidschendam
  - St. Antonius Ziekenhuis, Nieuwegein
  - Ikazia Ziekenhuis, Rotterdam
  - Antonius Ziekenhuis, Sneek
  - ZorgSaam Zeeuws Vlaanderen, Terneuzen
  - HAGA ziekenhuis, The Hague
  - ETZ, Tilburg
  - Diakonessenhuis, Utrecht
  - VieCuri Medisch Centrum, Venlo
  - Streekziekenhuis Koningin Beatrix (SKB), Winterswijk
  - Lange Land Ziekenhuis, Zoetermeer